CLINICAL TRIAL: NCT04011592
Title: Efficacy And Tolerability Of Sub-Anesthetic Ketamine In Postpartum Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment not feasible
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sudhakar Selvaraj, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-18-0416
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2020-09-14 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine 0.5 mg/kg, then Ketamine 0.2 mg/kg (Experimental): single intravenous infusion of Ketamine (0.5 mg/kg), washout period of seven days, and then single intravenous infusion of Ketamine (0.2 mg/kg)
  Interventions: Drug: Ketamine 0.5 mg/kg; Drug: Ketamine 0.2 mg/kg
- Ketamine 0.2 mg/kg, then Ketamine 0.5 mg/kg (Experimental): single intravenous infusion of Ketamine (0.2 mg/kg), washout period of seven days, and then single intravenous infusion of Ketamine (0.5 mg/kg)
  Interventions: Drug: Ketamine 0.5 mg/kg; Drug: Ketamine 0.2 mg/kg

INTERVENTIONS:
Drug: Ketamine 0.5 mg/kg — single intravenous infusion of Ketamine (0.5 mg/kg)
  Other Names: Ketamine Hydrochloride
Drug: Ketamine 0.2 mg/kg — single intravenous infusion of Ketamine (0.2 mg/kg)

SUMMARY:
Postpartum depression is a non-psychotic major or minor depressive episode that occurs during pregnancy or within 12 months of post-partum period. The nature of symptoms is same as depressive episode characterized by depressed mood, anxiety, sleep difficulties, suicidal thoughts, tiredness and diminished interest in pleasurable activities. Severe maternal depression affects children by increasing the risk of emotional and behavioral and physical health problems and cognitive difficulties. Thus early screening and intervention is critical in reducing the negative impact of PND in the mother and child, family and the community.

The purpose of this study is to assess the safety, pharmacokinetics and antidepressant efficacy of sub-anesthetic dose of intravenous ketamine in perinatal depression.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, ages 18-45 years
* Experienced a major depressive episode in the postpartum period beginning within the first 4 weeks following delivery and with moderate or severe symptoms (>12 EPDS or >14 HAM-D).
* No or partial response to adequate doses of SSRI medications to treat PND for longer than 6 weeks.
* PND patients will be requested to maintain the stable dose of antidepressants while enrolled in the study trial.
* Patients that can speak and read the English language, are able to understand the study procedures and sign the informed consent

Exclusion Criteria:

* No current or past psychosis or severe personality disorder.
* No current substance abuse or dependence.
* No serious and imminent suicidal or homicidal risk.
* No recent or history of major and unstable medical problems that affect brain anatomy, neurochemistry, or function.
* Not diagnosed with cardiovascular disorders.
* No increased risk of laryngospasm or active upper respiratory infections.
* Not diagnosed with an intellectual disability or neurodegenerative diseases.
* Mothers that are currently breastfeeding.
* No current pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Selvaraj, 713-486-2837, Principal Investigator — UTHealth Science Center at Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine 0.5 mg/kg, Then Ketamine 0.2 mg/kg | Ketamine 0.2 mg/kg, Then Ketamine 0.5 mg/kg
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one participant was enrolled, and this participant received 0.5 mg/kg Ketamine, then 0.2 mg/kg Ketamine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine 0.5 mg/kg, Then Ketamine 0.2 mg/kg | Ketamine 0.2 mg/kg, Then Ketamine 0.5 mg/kg | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (NA) — Standard Deviation is not calculable for 1 participant. |  | 37 (NA) — Standard Deviation is not calculable for 1 participant.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressed Mood as Indicated by Hamilton Depression Rating Scale (HAM-D) Score
Description: The Hamilton Depression Rating Scale (HAM-D) score ranges from 0-53. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity of depressive symptoms. The value reported is the score at baseline minus the score 24 hours post-injection.
Time Frame: baseline, 24 hours post-injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
Number analyzed (Participants) | 1 | 1
score on a scale | 9 (NA) — Standard Deviation is not calculable for 1 participant. | 3 (NA) — Standard Deviation is not calculable for 1 participant.

2. Secondary Outcome: Number of Treatment-Emergent Adverse Events
Time Frame: 24 hours post-injection
Measure: Number; unit: adverse events
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
Number analyzed (Participants) | 1 | 1
adverse events
  mild headache | 1 | 1
  moderate nausea | 1 | 0

3. Secondary Outcome: Change in Postnatal Depression as Indicated by Edinburgh Postnatal Depression Scale (EPDS) Scale
Description: The Edinburgh Postnatal Depression Scale (EPDS) score ranges from 0 to 30. Higher scores indicate worse outcome, with a score of 10 or greater indicating depression. The value reported is the score at baseline minus the score at 24 hours post-injection.
Time Frame: baseline, 24 hours post-injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
Number analyzed (Participants) | 1 | 1
score on a scale | 8 (NA) — Standard Deviation is not calculable for 1 participant. | 2 (NA) — Standard Deviation is not calculable for 1 participant.

4. Secondary Outcome: Change in Anxiety as Indicated by Generalized Anxiety Disorder 7-Item (GAD-7) Scale
Description: The Generalized Anxiety Disorder 7-Item (GAD-7) Scale score ranges from 0 to 21, with higher scores indicating greater anxiety. The value reported is the score at baseline minus the score 24 hours post-injection.
Time Frame: baseline, 24 hours post-injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
Number analyzed (Participants) | 1 | 1
score on a scale | 5 (NA) — Standard Deviation is not calculable for 1 participant. | 0 (NA) — Standard Deviation is not calculable for 1 participant.

5. Secondary Outcome: Change in Depression as Indicated by Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) score ranges from 0 to 27, with greater scores indicating more severe depression.
Time Frame: baseline, 24 hours post-injection
Population: This outcome measure was not assessed and no data were collected.
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Behavioral Suicidal Events (Suicidal Ideation), as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a suicidal ideation and behavior rating scale with yes/no responses. The first part (Items 1-5) rates an individual's degree of suicidal ideation on a 0-5 scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent and behaviors". The C-SSRS outcomes are categories and have binary responses (yes/no). Suicidal ideation is considered when the patient responds a "yes" answer at any time during treatment to any one of the five suicidal ideation questions (Categories 1-5) on the C-SSRS. The sum of the 5 intensity item scores create a total score (range 0 to 25) to represent the intensity rating (higher scores indicate more severe suicidal ideation).
Time Frame: baseline, 24 hours post-injection
Population: This outcome measure was not assessed and no data were collected.
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Behavioral Suicidal Events (Suicidal Behavior), as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The questions 6-10 of the C-SSRS are related to suicidal behavior, and the outcome is a simple yes/no response. Suicidal behavior occurs if the patient answers a "yes" at any time during treatment to any one of the five suicidal behavior questions (Categories 6-10) on the C-SSRS.
Time Frame: baseline, 24 hours post-injection
Population: This outcome measure was not assessed and no data were collected.
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Ketamine 0.5 mg/kg | Ketamine 0.2 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.5 mg/kg (N=1) | Ketamine 0.2 mg/kg (N=1)
Mild headache (General disorders) | 1 (1) | 1 (1)
Moderate Nausea (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Only one subject was enrolled, and enrollment goal not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT04011592/Prot_SAP_000.pdf